CLINICAL TRIAL: NCT02983175
Title: Ultrasound Assessment of Gastric Content and Gastric Volume Before Crash Induction for Appendectomy
Brief Title: Ultrasound Assessment of Gastric Content Before Anesthesia for Appendectomy
Acronym: EGASTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-A01501-50
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Appendectomy
Keywords: ultrasonogaphy; full stomach; pulmonary aspiration; anaesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasound assessment of gastric content (Experimental)
  Interventions: Other: ultrasound assessment of gastric content

INTERVENTIONS:
Other: ultrasound assessment of gastric content — Achievement of gastric ultrasound (specific procedure) :
  Gastric ultrasound is performed specifically for the study by a senior anesthetist physician in a patient placed supine, semi-sitting by an angle of 45 ° relative to the horizontal.
  Standardised achievement of the antral ultrasound by the following method:
  * First, a qualitative assessment of antral contents in 3 grades according to the "Perlas" method [24].
  * Second, performing a quantitative analysis of antral contents calculating the CSA.
  * Then, volume of gastric contents calculation as from the CSA.

SUMMARY:
Performing anesthetic induction for appendicectomy has two main risks : first aspiraion of gastric content causing pneumonia. Otherwise, anaphylactic risk to drugs used during anesthetic induction. Indeed, the guidelines recommend an anesthetic induction protocol qualified "full stomach" whatever the patient and the preoperative fasting period are. This protocol provides the use of fast-acting neuromuscular blocking agents (succinylcholine or rocuronium). However, these neuromuscular blocking agents are ten times more at allergic risk than others. Ultrasound assessment of gastric content before rapid sequence induction of anesthesia is a reproducible, non-invasive, inexpensive and quickly achievable bedside technique. Furthermore, the correlations between gastric volume and risk of a full stomach and also between the cross-section antral area (CSA) and the risk of a full stomach have been validated on several patient cohorts. We formulate the hypothesis that the achievement of a gastric ultrasound before anesthetic induction for appendectomy could allow to identify "full stomach" patients who actually justify rapid sequence induction of anesthesia with exposure to fast-acting neuromuscular blocking agents that implies.

Primary endpoint is to determine te percentage of patients who have a gastric content before appendectomy. Secondary endpoint is to determine the incidenc of aspiration pneumonia and anaphylactic shock. Another secondary endpoint is to determine the percentage of patient with gastric content with the antral grading system (Perlas method) and to evaluate the concordance between this methode and the cross-section antral area.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the operating room for appendectomy.
* Major or minor patient (higher than 16) affiliated to a social security scheme.
* Patient or parents of minor patient who received the full information relative to the organization of the study and who signed his/their informed consent(s).

Exclusion Criteria:

* Pregnant women.
* Childbearing age patient does not have effective contraception.
* Breastfeeding woman.
* Minor patient under 16.
* Major patient subject to a measure of legal protection or unable to consent.
* Persons deprived of liberty by a judicial or an administrative decision.
* Patient with gastric and/or esophagus surgery history.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Cross-section antral area (CSA) | baseline J0
  Ultrasonography exam of the stomach is used to evaluate the CSA. A CSA greater than 340mm² defines a full stomach. The calculation of the CSA is : CSA = AP x CC x π / 4 (in mm²). With AP - antero-posterior gastric antrum diameter and CC - cranio-caudal gastric antrum diameter

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bouvet L, Mazoit JX, Chassard D, Allaouchiche B, Boselli E, Benhamou D. Clinical assessment of the ultrasonographic measurement of antral area for estimating preoperative gastric content and volume. Anesthesiology. 2011 May;114(5):1086-92. doi: 10.1097/ALN.0b013e31820dee48. PMID 21364462
- [Result] Perlas A, Chan VW, Lupu CM, Mitsakakis N, Hanbidge A. Ultrasound assessment of gastric content and volume. Anesthesiology. 2009 Jul;111(1):82-9. doi: 10.1097/ALN.0b013e3181a97250. PMID 19512861
- [Result] Reddy JI, Cooke PJ, van Schalkwyk JM, Hannam JA, Fitzharris P, Mitchell SJ. Anaphylaxis is more common with rocuronium and succinylcholine than with atracurium. Anesthesiology. 2015 Jan;122(1):39-45. doi: 10.1097/ALN.0000000000000512. PMID 25405395